CLINICAL TRIAL: NCT07145021
Title: The Effects of Breathing Exercises Administered to Associate Degree Students on Test Anxiety and Academic Achievement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Minel YILDIRIM, Lecturer, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ISTANBUL MEDIPOL UNIVERSITY
Record Dates: First submitted 2025-08-10; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Breath Exercise; Test Anxiety; Higher Education Students; Academic Achievement
Keywords: Breathing exercises, test anxiety, academic achievement, associate degree students, stress management, higher education

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing Exercise Intervention Group (Active Comparator)
  Interventions: Behavioral: Breathing Exercise Intervention
- Control Group (No Intervention) (No Intervention)

INTERVENTIONS:
Behavioral: Breathing Exercise Intervention — Participants will receive guided breathing exercise training conducted by a certified breathing coach. The intervention consists of weekly 40-minute sessions over a 6-week period, aimed at reducing test anxiety and improving academic performance. Participants will also maintain a breathing exercise log throughout the study.
  Arms: Breathing Exercise Intervention Group

SUMMARY:
This study aims to examine the effects of breathing exercises administered to associate degree students on test anxiety and academic achievement.

Primary Research Question:

Do breathing exercises administered to associate degree students reduce test anxiety and improve academic achievement?

Researchers will compare the effects of breathing exercises on test anxiety and academic achievement by using a control group (no breathing exercise intervention) and an intervention group.

Participants:

All students from a vocational school who consent to participate will be administered the Westside Test Anxiety Scale.

Students with high anxiety scores will be assigned to the intervention group.

The intervention group will receive breathing exercise training delivered by a certified Breathing Coach (the researcher).

Breathing exercises will be conducted for 40 minutes per week, over a 6-week period.

Students will be asked to maintain a breathing exercise log.

Following the end-of-term examinations, data collection forms will be re-administered and results will be compared between pre- and post-intervention assessments.

DETAILED DESCRIPTION:
This study aims to investigate whether breathing exercises can help reduce test anxiety and improve academic performance in undergraduate students. Students who volunteer will complete a short test anxiety questionnaire. Those with higher levels of test anxiety will be randomly assigned to an intervention group or a control group. The intervention group will practice breathing exercises once a week for 45 minutes over 8 weeks and receive information on coping strategies for test anxiety. The study will examine changes in test anxiety and course exam scores.

ELIGIBILITY:
Inclusion Criteria:

* Vocational school students
* Obtaining informed consent from students
* No language, hearing, intellectual, or psychological impairments
* Ability to speak and understand Turkish
* Willingness to participate in the study

Exclusion Criteria:

* Presence of any chronic disease
* Use of any psychiatric medication

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-22 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Test Anxiety Scores as measured by the Westside Test Anxiety Scale (WTAS) | 6 months
  The Westside Test Anxiety Scale (WTAS) will be administered to all students who volunteer to participate in the study. Students with scores one point above the mean or higher will be considered to have high test anxiety. Those identified as having high anxiety will be randomized into intervention and control groups. The intervention group will receive breathing exercises once per week for 45 minutes over a period of 8 weeks, in addition to receiving information about test anxiety and coping strategies. Breathing exercises, such as the 4-4-4-4 technique and the 4-7-8 technique, will be taught and practiced with the students.
End-of-Term Course Exam Score (%) | 6 months
  Academic performance will be evaluated using the official end-of-term course exam score reported by the institution (0-100%). The outcome will be summarized as the mean score at Week 8 and between-group difference.

SECONDARY OUTCOMES:
Adherence to Breathing Exercise Intervention (% of Planned Sessions Attended) | 6 Month
  For students in the intervention group, adherence to the breathing exercise program will be calculated as the percentage of scheduled sessions attended. A total of 8 sessions, once per week for 45 minutes, will be offered. The mean attendance rate and distribution across participants will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Minel YILDIRIM, Principal Investigator

IPD SHARING:
Plan to Share IPD: No